CLINICAL TRIAL: NCT06203990
Title: Barre Exercise for People With Parkinson Disease
Brief Title: Barre Exercise in Parkinson's
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gammon M Earhart, Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202312097
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Barre class (Experimental): Barre is an exercise modality that combines elements of classical ballet with strength training. Barre involves high repetitions of low impact, isometric movements, requires little to no equipment, and is highly modifiable for different fitness levels. Barre is traditionally performed in a class setting, which promotes increased social interaction and builds community. Furthermore, interventions with dance elements exhibit high adherence rates (often > 80%).The exercises in a barre class are also performed holding on to a fixed barre or on the floor, which may address people with PD's fear of falling.
  Interventions: Behavioral: Barre exercise

INTERVENTIONS:
Behavioral: Barre exercise — Group barre exercise class

SUMMARY:
This study asks if a barre exercise program is a feasible and acceptable form of exercise for individuals with Parkinson disease. The study will also evaluate barre's potential effects on motor outcomes, including balance, strength, and functional mobility.

DETAILED DESCRIPTION:
The primary objectives of this study are to: 1) evaluate the feasibility and acceptability of a barre exercise intervention and 2) gather preliminary data regarding the effect of a barre exercise intervention on balance, strength, functional mobility and quality of life in individuals with mild to moderate Parkinson disease (PD). Individuals with PD (N=15) will be recruited to participate in a pilot barre exercise class led by a certified barre instructor. The intervention will include 24, 45-50 minute group classes (twice weekly for 12 weeks, excluding holidays). Pre- and post-intervention data collection will include assessments of balance, lower extremity strength, and functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by a neurologist with idiopathic Parkinson disease
* at least 18 years of age
* a score on the Hoehn & Yahr (H&Y) scale between I-III to indicate mild to moderate disease severity
* able to provide informed consent
* able to walk for 10 continuous minutes without assistance from another person
* stable medication regimen for at least one month prior to enrollment

Exclusion Criteria:

* any neurological condition other than PD
* history of orthopedic or other medical conditions that limit the ability to safely participate in the intervention or
* language, visual, or hearing barriers to participation
* evidence of dementia (Montreal Cognitive Assessment < 24) to ensure understanding of the intervention class instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2024-February 2024, Participants recruited from an academic medical center
Pre-assignment Details: No significant events occurred after participant enrollment. Participants were only enrolled if they met inclusion criteria.
Period: Overall Study
Arm/Group | Barre Class
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Barre Class
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Movement Disorders Society Unified Parkinson Disease Rating Scale Part III (MDS-UPDRS-III) [Mean (Standard Deviation); unit: scores on a scale] — MDS-UPDRS Part III: Motor Examination. A measure of Parkinson disease motor symptom severity rated on a scale from 0-132. Higher scores indicate more severe motor impairment, reflecting a worsening of symptom severity.
  scores on a scale | 26 (5)

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: Number of participants who attended at least 75% of the classes
Time Frame: 12 weeks
Population: Two participants withdrew from the study during the intervention period. Attendance was calculated for the 11 participants who remained enrolled for the duration of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Barre Class
Number analyzed (Participants) | 11
Participants | 10

2. Primary Outcome: Retention (Study Completion)
Description: Percent of participants who remained enrolled for the duration of the study
Time Frame: 12 weeks
Population: Thirteen participants enrolled in the classes. Two participants withdrew from the study during the intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Barre Class
Number analyzed (Participants) | 13
Participants | 11

3. Secondary Outcome: Balance
Description: Mean change in total score on the Mini Balance Evaluation Systems Test (Mini-BESTest) from pre- to post-intervention. The Mini-BESTest is a brief, clinically relevant assessment of balance, scored on a scale from 0 to 28, with higher scores indicating better balance. A negative change score reflects a decline in balance performance from pre- to post-intervention.
Time Frame: 12 weeks
Population: Two participants withdrew from the study during the intervention period. Following the intervention, one participant was not able to return for in-person balance assessment and one participant was excluded from preliminary motor trend data due to severe freezing of gait. Nine participants were analyzed for preliminary motor trends.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Barre Class
Number analyzed (Participants) | 9
scores on a scale | -0.67 (1.58)

4. Secondary Outcome: Functional Strength
Description: Mean change in time taken to complete five sit to stand movements pre- to post- intervention, measured in seconds. Longer time indicates worse performance.
Time Frame: 12 weeks
Population: Two participants withdrew from the study during the intervention period. Following the intervention, one participant was not able to return for in-person functional strength assessment and one participant was excluded from preliminary motor trend data due to severe freezing of gait. Nine participants were analyzed for preliminary motor trends.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Barre Class
Number analyzed (Participants) | 9
seconds | 1.45 (3.10)

5. Secondary Outcome: Gait
Description: Mean change in gait speed pre- to post-intervention, measured in meters/second.
Time Frame: 12 weeks
Population: Two participants withdrew from the study during the intervention period. Following the intervention, one participant was not able to return for in-person gait assessment and one participant was excluded from preliminary motor trend data due to severe freezing of gait. Nine participants were analyzed for preliminary motor trends.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Barre Class
Number analyzed (Participants) | 9
m/s | 0.05 (0.08)

6. Primary Outcome: Acceptability
Description: Mean group rating on the Client Satisfaction Questionnaire, a standardized measure using Likert-scale questions to assess self-reported satisfaction of a program. Range is 1-4, higher scores indicate higher satisfaction
Time Frame: 12 weeks
Population: All participants who completed the intervention completed the client satisfaction questionnaire.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Barre Class
Number analyzed (Participants) | 11
scores on a scale | 3.8 [3 to 4]

ADVERSE EVENTS:
Time Frame: From enrollment until end of post-testing, up to 17 weeks.
Description: An adverse event is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical or clinical treatment or procedure that may or may not be considered related to the medical or clinical treatment or procedure.
Arm/Group | Barre Class
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Barre Class (N=13)
Fall (Musculoskeletal and connective tissue disorders) | 2 (4) — Mild Grade 1, events unrelated to intervention
Fall (Musculoskeletal and connective tissue disorders) | 4 (4) — Moderate Grade 2, events unrelated to intervention
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Moderate Grade 2, reasonable possibility related to invention, reported lower back pain prior to enrolling in the study
Dizziness Due to Low Blood Pressure (Cardiac disorders) | 1 (1) — Mild Grade 1, unrelated to intervention
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Severe Grade 3, unrelated to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT06203990/Prot_SAP_000.pdf